CLINICAL TRIAL: NCT02167477
Title: Comparison of the C-MAC Video Laryngoscope With Conventional Direct Laryngoscopy in Morbidly Obese Patients Using a Photographic Overlay Technique
Brief Title: Comparison of Indirect and Direct Laryngoscopy in Obese Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/NW/0805
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2016-03

CONDITIONS: OBESITY, MORBID; BARIATRIC SURGERY CANDIDATE
Keywords: Intubation, Endotracheal
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngoscopy sequence 1 (Active Comparator): Macintosh laryngoscopy Storz C-MAC, standard blade Storz C-MAC, D-BLADE
  Interventions: Device: Macintosh laryngoscopy; Device: Storz C-MAC, standard blade; Device: Storz C-MAC, D-BLADE
- Laryngoscopy sequence 2 (Active Comparator): Macintosh Storz C-MAC, D-BLADE Storz C-MAC, standard blade
  Interventions: Device: Macintosh laryngoscopy; Device: Storz C-MAC, standard blade; Device: Storz C-MAC, D-BLADE

INTERVENTIONS:
Device: Macintosh laryngoscopy — Tracheal intubation
Device: Storz C-MAC, standard blade — Tracheal intubation
Device: Storz C-MAC, D-BLADE — Tracheal intubation

SUMMARY:
An anaesthetist inserts a "laryngoscope" into the mouth to see the voice-box (larynx) for "tracheal intubation", when a tube is advanced into the windpipe (trachea) to protect the airway and administer anaesthetic gases.

This study aims to compare traditional (direct view) Macintosh (MAC) laryngoscopy with Storz C-MAC videolaryngoscopes in subjects presenting for obesity reduction surgery using a novel "photographic overlay technique" to analyse the basis for any differences.

DETAILED DESCRIPTION:
The aim is to have 40 patients complete the protocol. This number is based on a recent similar study at Aintree hospital where this number of cases was successfully used to make multiple parameter comparisons between different videolaryngoscope blades during Ear Nose and Throat (ENT) procedures. Following the template of this earlier work all the patients will have three laryngoscopy assessments.

When seen in the preoperative clinic, patients will be informed about the study and given a patient information sheet to take home. On the day of admission for surgery they will be asked for their consent to be involved in the study by the study researchers.

Prior to theatre, the research team will make a number of straightforward external measurements. Various surface markings around the head and neck of the patients will be applied immediately before proceeding to the operating theatre. In the anaesthetic room, prior to induction of anaesthesia, the patients will have standard monitoring attached (including oxygen saturations, electrocardiograph and non-invasive blood pressure). They will be positioned as usual by the anaesthetist in charge of the case. The monitoring of the laryngoscopy will comprise:

1. Video-camera recording one metre away from the side of the patient's head and neck.
2. Photographic still shots at the moment of laryngoscopy from the foot of the bed/trolley.
3. View of laryngoscopy itself via the optical systems in the C-MAC® video laryngoscopes The photographs taken from the foot of the bed/trolley are to note any lateral rotation in the head position during laryngoscopy. Should this occur it may need to be allowed for in the processing of the photographic overlay analysis during processing of the lateral images.

The anaesthetic technique will be standardised. After 3 mins of pre-oxygenation with a face mask, anaesthesia is induced with Remifentanil (technique for administration will be decided by the individual anaesthetist), Propofol 1.5-2.5 mg/kg and neuromuscular blockade with Rocuronium 0.6 mg/kg before airway manipulation. Bag mask ventilation with 100% oxygen and volatile anaesthetic will be performed prior to and between each of the three laryngoscopy assessments. The patient will be monitored closely for any adverse signs, if at any point the oxygen saturations fall below 90% the patient will be withdrawn from the study and anaesthesia continued as deemed appropriate by the responsible clinician. During each laryngoscopy the anaesthetist will indicate when the moment of maximal laryngoscopic view is obtained so that this can be recorded by the video devices. In the case of Macintosh, the observed percentage of glottic opening or POGO score will be documented. If an inadequate view is found the clinician may have one attempt at improving the view with cricoid pressure which will again be recorded. The conventional Macintosh laryngoscope will always be used for the first laryngoscopy. The sequence of the second and third laryngoscopies will be decided by block randomisation. Tracheal intubation will be undertaken during the final laryngoscopy. A shaped metallic stylet will be place within the tracheal tube as an intubation aid in all patients intubated with the C-MAC® D-BLADE video laryngoscope. Following intubation, an endoscopic examination of the posterior wall of the pharynx will be undertaken as the videolaryngoscope is withdrawn to ensure no trauma has been caused by the intubation. Following intubation, the patient will then continue with anaesthesia and surgery as planned. There will be monitoring of the patient closely in recovery and post-operatively as part of normal clinical care.

Off-line data analysis will consist of superposition of the videolaryngoscope blade shape outlines on the lateral photographic images. The POGO scores will be compared with the preoperative measurements and the relevant results from the overlay imaging analysis.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (BMI >35) for elective bariatric surgery

Exclusion Criteria:

* Patients in whom rapid sequence induction of anaesthesia is indicated
* Patients in whom the responsible anaesthetist considers conventional laryngoscopy inappropriate (e.g. when the mouth opening is too narrow)
* Patients whose comorbidity makes them unsuitable for this type of study (e.g. those with limited cardiopulmonary reserve)
* patients who do not consent to be involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
POGO (percentage of glottic opening) score at maximum laryngeal view for three laryngoscopes (Macintosh, Storz C-MAC, standard and D-BLADE) | one year

SECONDARY OUTCOMES:
Subjective "ease of intubation" | one year
Time to intubate | one year

OTHER OUTCOMES:
Anatomical features important in ensuring an adequate view of the larynx | one year
Differences in what ensures an adequate view of the larynx for direct and indirect viewing devices | one year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Charters, Principal Investigator — Aintree University Hospitals
Locations (1):
- Aintree University Hospitals, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charters P. Analysis of mathematical model for osseous factors in difficult intubation. Can J Anaesth. 1994 Jul;41(7):594-602. doi: 10.1007/BF03009999. PMID 8087908